CLINICAL TRIAL: NCT03699956
Title: A Phase 3, Controlled, Open-label, Randomized Study of RRx-001 Administered Sequentially With a Platinum Doublet or a Platinum Doublet in Third-Line or Beyond Small Cell Lung Cancer
Brief Title: RRx-001 Sequentially With a Platinum Doublet or a Platinum Doublet in Third-Line or Beyond in Patients With Small Cell Lung Cancer
Acronym: REPLATINUM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: RRx-001 will be studied under a new global, phase 3 clinical trial
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-33
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Carcinoma, Small Cell Lung
Keywords: RRx-001; Lung Cancer; Lung Neoplasms; Phase 3; Immunotherapy; Small Cell Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms; Carcinoma, Small Cell | interventions — RRx-001; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Intervention Model Description: In this study, patients will be randomized to 1 of 2 groups or arms. Patients in Arm 1 will receive the study drug, RRx-001, once a week for 3 weeks followed by up to 4 cycles of platinum doublet (platinum plus etoposide) chemotherapy. Patients with stable disease or better will go on to the Platinum Stacking Phase and will receive RRx-001 once a week for 2 weeks followed by 2 cycles of single agent platinum chemotherapy in a repeating pattern until such time as their cancer gets worse.. Patients in Arm 2 will receive the standard of care platinum doublet (platinum plus etoposide) chemotherapy for up to 4 cycles. . Patients in arm 2 whose cancer gets worse (as determined by imaging scans), may "cross-over" to the Platinum Stacking Phase of Arm 1 (see study schema below).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): RRx-001 + eLOOP Device 4 mg IV infusion once weekly for 3 weeks
  Cisplatin/carboplatin plus etoposide (up to 4 cycles):
  1. Cisplatin or Carboplatin:
     1. Cisplatin initially dosed at 60 mg/m2 on Day 1 every 3 weeks OR
     2. Carboplatin initially dosed at an AUC (area under the curve) of 5 on Day 1 every 3 weeks
  2. Etoposide to be given per the initial approval by the package insert (USPI FDA) at 100 mg/m2 Days 1-3 every 3 weeks
  Interventions: Combination Product: RRx-001 + eLOOP Device; Drug: Cisplatin/carboplatin plus etoposide
- Arm 2 (Active Comparator): Cisplatin/carboplatin plus etoposide (up to 4 cycles):
  1. Cisplatin or Carboplatin:
     1. Cisplatin initially dosed at 60 mg/m2 on Day 1 every 3 weeks OR
     2. Carboplatin initially dosed at an AUC of 5 on Day 1 every 3 weeks
  2. Etoposide to be given per the initial approval by the package insert (USPI FDA) at 100 mg/m2 Days 1-3 every 3 weeks
  Interventions: Drug: Cisplatin/carboplatin plus etoposide

INTERVENTIONS:
Combination Product: RRx-001 + eLOOP Device — RRx-001 is a small molecule anticancer drug which is mixed with patient's own blood using the eLOOP device
  Arms: Arm 1
Drug: Cisplatin/carboplatin plus etoposide — Standard of care platinum doublet chemotherapy

SUMMARY:
This Phase 3 study aims to find out whether RRx-001 + platinum chemotherapy is more effective than platinum chemotherapy alone in 3rd line or beyond small cell cancer.

DETAILED DESCRIPTION:
Small cell cancer (SCC), which mostly arises in the lungs but also in other parts of the body as well such as the prostate and the intestines, is one of the most aggressive forms of cancer; in fact, SCC is so aggressive that in 2012 Congress designated it a recalcitrant or difficult-to-treat cancer, along with pancreatic cancer and glioblastoma or GBM, a primary tumor of the brain, which share the terrible "distinction" of having a 5 year survival rate less than 50%.

One of the main reasons that SCC is so recalcitrant or difficult-to-treat has to do with the development of resistance. Almost all cancers (and SCC is no exception) are treated according to lines of therapy. A line of therapy is a particular course of treatment or treatment regimen. So, in SCC, the first line of treatment is a platinum doublet, with the word doublet meaning two, and consists of the double chemotherapy regimen of cisplatin or carboplatin + etoposide. Most patients initially respond well to the platinum doublet but unavoidably, as a matter of course, resistance to treatment develops and, with that development, a new treatment in second line is started. The same pattern is followed in later lines of therapy: resistance in second line leads to the start of another treatment in 3rd line, and with resistance in 3rd line, which is, unfortunately, just as inevitable, and usually happens even sooner, since the later the line of therapy the more aggressive the tumor, a 4th line treatment is started and so on and so forth until, eventually, no lines of treatment are left. The implicit or unwritten rule in cancer therapy is that once resistance occurs on a particular treatment that same treatment is never reintroduced or restarted.

RRx-001 is a form of immunotherapy that has the potential to overturn this unwritten rule by sensitizing tumors, in other words, by making them more sensitive to the platinum doublet that they received in first line. This is very important because, as previously stated, the platinum doublet is usually the most effective therapy, so it is a benefit to patients if sensitivity to the platinum doublet is restored or increased (even in cases where no response ever occurred) and now they respond as if they were in 1st line rather than in 3rd line or beyond.

In this study, which is called REPLATINUM, because patients will be reintroduced to or restarted on a platinum doublet, there is a 50% chance of receiving either RRx-001 + platinum doublet in Arm 1 or a platinum doublet without RRx-001 in Arm 2. However, patients in arm 2 whose cancer progresses or gets worse (as determined by imaging scans), have the opportunity to "cross-over" to Arm 1 and receive RRx-001 + platinum doublet until such time as their cancer progresses. In this way, all patients, even those on Arm 2, are potentially eligible to be treated with RRx-001.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and < 80 years
2. Prior platinum treatment is required
3. Prior treatment with a checkpoint inhibitor is required unless contraindicated. Maintenance with a checkpoint inhibitor is NOT required
4. Patient must have received at least 2 prior lines of therapy
5. Biopsy confirmation of small cell lung cancer
6. Capable of providing informed consent and complying with trial procedures
7. Measurable disease by RECIST 1.1. Measurable lesions will be confirmed by imaging (CT scan)
8. PS 0-1

Exclusion Criteria:

1. Symptomatic central nervous system metastases or neurologically unstable patients that are on increasing steroid dose.
2. The presence of another primary malignancy (excluding in situ of the cervix or basal carcinoma of the skin)
3. Treatment of SCLC with any antineoplastic agent with the exception of steroids.
4. Patients with clinically significant illnesses which would compromise participation in the study, including, but not limited to active or uncontrolled infection, immune deficiencies, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, certain heart conditions, or mental illness/social situations that would limit compliance with study requirements.
5. History of an allergic reaction to previously received platinum-based regimen, or history of having to discontinue previously received platinum-based regimen secondary to toxicity (excluding hematologic toxicity)
6. Any clinical laboratory findings, which give reasonable suspicion of a disease or condition that contraindicates the use of any study medication or renders the patient at high risk from treatment
7. Uncontrolled or symptomatic pleural or pericardial effusion
8. Pregnant or nursing. There is a potential for congenital abnormalities and for this regimen to harm nursing infants

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Estimated up to 12 Months
  The time from the date of randomization to disease progression (radiologic and/or symptomatic per RECIST 1.1) or death from any cause

SECONDARY OUTCOMES:
Overall Survival | Estimated up to 12 Months
  The time from randomization to death from any cause
Overall response rate | Estimated up to 12 Months
  The proportion of patients with a complete response or a partial response (per RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Oronsky, MD, PhD, Study Director — EpicentRx, Inc.
Locations (18):
- United States (18):
  - Centura Health Research Center, Denver, Colorado
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - AdventHealth Hematology and Oncology, Orlando, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Cotton O'Neil Clinical Research Center.Hematology & Oncology, Topeka, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - University of Maryland Marlene and Stewart Greenbaum Comprehensive Cancer Center, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Millennium Oncology, Houston, Texas
  - HOPE Cancer Center of East Texas, Tyler, Texas
  - Utah Cancer Specialist, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jayabalan N, Oronsky B, Cabrales P, Reid T, Caroen S, Johnson AM, Birch NA, O'Sullivan JD, Gordon R. A Review of RRx-001: A Late-Stage Multi-Indication Inhibitor of NLRP3 Activation and Chronic Inflammation. Drugs. 2023 Apr;83(5):389-402. doi: 10.1007/s40265-023-01838-z. Epub 2023 Mar 15. PMID 36920652
- [Derived] Oronsky B, Reid TR, Larson C, Caroen S, Quinn M, Burbano E, Varner G, Thilagar B, Brown B, Coyle A, Ferry L, Abrouk N, Oronsky A, Scribner CL, Carter CA. REPLATINUM Phase III randomized study: RRx-001 + platinum doublet versus platinum doublet in third-line small cell lung cancer. Future Oncol. 2019 Oct;15(30):3427-3433. doi: 10.2217/fon-2019-0317. Epub 2019 Sep 11. PMID 31509028